CLINICAL TRIAL: NCT06787170
Title: Prediction of Platinum Resistance and Prognosis in Patients with High-grade Serous Ovarian Cancer Based on MRI Habitat Imaging and Radiopathomics
Brief Title: Prediction of Platinum Resistance and Prognosis of High-grade Serous Ovarian Cancer
Acronym: PPRPHGSOC
Status: Completed | Type: Observational
Sponsor: The First People's Hospital of Yunnan (Other)
Responsible Party: Principal Investigator, Qiu Bi, Dr., The First People's Hospital of Yunnan
Other Study IDs: KHLL2023-KY208; 82460340 (Other Grant/Funding Number: National Natural Science Foundations of China)
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: High-grade Serous Ovarian Cancer (HGSOC)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: MRI habitat imaging — Habitat imaging, a data-driven image processing technique that divides the entire lesion into multiple sub-regions without assuming anything prior, has capacity to noninvasively evaluate the intratumoral heterogeneity.
  Other Names: radiopathomics

SUMMARY:
High-grade serous ovarian carcinoma (HGSOC) is the most common subtype of ovarian carcinoma. Platinum-based drugs are the first-line chemotherapeutic agents for HGSOC, but platinum resistance and prognosis are difficult to predict. Domestic and foreign studies have found that multi-functional MRI could reflect the macroscopic heterogeneity of tumors from different perspectives; habitat imaging contributed to reflecting the spatial heterogeneity of tumors; the attention mechanism could integrate features of different scales; and multi-omics were capable to improve predictive performance. Previously, our team has demonstrated the importance of MRI and its functional imaging in the diagnosis and histological evaluation of gynecological tumors. And conventional MRI habitat imaging, multi-instance learning based on whole slide image (WSI), and multi-omics model could effectively predict platinum resistance in HGSOC patients. Therefore, this study aims to perform habitat imaging on multi-functional MRI such as multi b-value DWI and DCE-MRI and to train WSI-based multi-instance learning to construct pathological signature. Then, combined with clinical indicators, radiomics based on MRI habitat, and pathomics, a multi-omics fusion model trained by attention mechanism was constructed. Finally, to explore the value of MRI habitat, WSI, and multi-omics in predicting platinum resistance and prognosis in HGSOC patients. This study combines macroscopic functional imaging and microscopic pathological information to construct a multi-omics complementary model, which can predict platinum resistance and prognosis of HGSOC patients more comprehensively and accurately, and further guide the formulation of clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as HGSOC based on surgery and pathology.
* The standard treatment including surgical cytoreduction followed by at least three cycles of regular platinum-based chemotherapy after surgery.
* Follow-up records available for more than six months after postoperative chemotherapy.
* For MRI analysis, pelvic MRI examination including axial T2-weighted imaging (T2WI), contrast-enhanced T1-weighted imaging (CE-T1WI), and diffusion-weighted imaging (DWI) was performed within two weeks prior to treatment, and patients had no any treatments other than neoadjuvant chemotherapy (NACT) performed between MRI and surgery.

Exclusion Criteria:

* Patients with a history of platinum-based chemotherapy for other malignancies.
* Absence of essential clinical data.
* For MRI analysis, patients with poor MRI imaging quality and registration, or a tumor maximum diameter < 1 cm on MRI needed to be excluded.
* For pathology analysis, patients without H&E-stained WSIs or with poor WSI imaging quality should be excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HGSOC patients confirmed by surgery and pathology
Sampling Method: Non-Probability Sample
Enrollment: 1129 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
platinum resistance | within 6 months
  Platinum resistance is determined based on whether there is disease progression during or within 6 months after termination of platinum-based chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Bi, Principal Investigator — The First People's Hospital of Yunnan
Locations (1):
- the First People's Hospital of Yunnan Province, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No